CLINICAL TRIAL: NCT00990964
Title: Attain Success Clinical Trial
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Attain Success
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-08

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Attain Success Lead — Attain Success Lead

SUMMARY:
The purpose of the study is to assess lead implant success and complication rate using the Medtronic Attain Family of left-heart leads and delivery catheters.

ELIGIBILITY:
Inclusion Criteria:

* Subject is at least 18 years of age or older
* Subject will be implanted with Medtronic cardiac resynchronization therapy (CRT) device and Medtronic left heart lead utilizing (or attempting to utilize) Attain Family of delivery catheters. The implant procedure may include upgrades to CRT from implantable pulse generator (IPG) or implantable cardioverter-defibrillator (ICD).

Exclusion Criteria:

* Subject is enrolled in a concurrent study with the exception of a study approved by the Medtronic Clinical Trial Leader prior to enrollment
* Subject has existing CRT system implanted or was previously implanted with a CRT system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient referral to a participating study center with practitioners experienced in handling and implantation of the cardiac resynchronization therapy (CRT) device, the left-heart lead, and the use of the delivery catheter.
Sampling Method: Non-Probability Sample
Enrollment: 2014 (Actual)
Dates: Start 2009-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John D Hummel, MD, Principal Investigator — Davis Heart & Lung Research Institute, The Ohio State University
Locations (108):
- United States (72):
  - Little Rock, Arkansas
  - Downey, California
  - Modesto, California
  - Redding, California
  - Riverside, California
  - San Diego, California
  - San Jose, California
  - Santa Rosa, California
  - Danbury, Connecticut
  - Washington D.C., District of Columbia
  - Delray Beach, Florida
  - Lake Mary, Florida
  - Naples, Florida
  - Orlando, Florida
  - Panama City, Florida
  - Saint Augustine, Florida
  - Tampa, Florida
  - Athens, Georgia
  - Atlanta, Georgia
  - Macon, Georgia
  - Marietta, Georgia
  - Chicago, Illinois
  - Decatur, Illinois
  - Indianapolis, Indiana
  - Newburgh, Indiana
  - Overland Park, Kansas
  - Bowling Green, Kentucky
  - Lexington, Kentucky
  - Houma, Louisiana
  - Baltimore, Maryland
  - Takoma Park, Maryland
  - Boston, Massachusetts
  - Muskegon, Michigan
  - Royal Oak, Michigan
  - Saint Clair Shore, Michigan
  - Ypsilanti, Michigan
  - Minneapolis, Minnesota
  - St Louis, Missouri
  - Washington, Missouri
  - Omaha, Nebraska
  - Concord, New Hampshire
  - Englewood, New Jersey
  - Huntington, New York
  - Asheville, North Carolina
  - Concord, North Carolina
  - Fargo, North Dakota
  - Cleveland, Ohio
  - Columbus, Ohio
  - Kettering, Ohio
  - Abington, Pennsylvania
  - Bethlehem, Pennsylvania
  - Erie, Pennsylvania
  - Harrisburg, Pennsylvania
  - Wormleysburg, Pennsylvania
  - Florence, South Carolina
  - Germantown, Tennessee
  - Knoxsville, Tennessee
  - Nashville, Tennessee
  - Amarillo, Texas
  - Austin, Texas
  - Brownsville, Texas
  - Dallas, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Longview, Texas
  - The Woodlands, Texas
  - Murray, Utah
  - Salt Lake City, Utah
  - Frederickburg, Virginia
  - Bellingham, Washington
  - Spokane, Washington
  - Green Bay, Wisconsin
- Ontario, Canada
- China (3):
  - Jiangsu
  - Sichuan
  - Xinjian
- France (12):
  - Amiens
  - Anglouleme
  - Bayonne
  - Bordeaux
  - Clermont-Ferrand
  - Créteil
  - Metz-Tessy
  - Montfermeil
  - Nice
  - Orléans
  - Paris
  - Poitiers
- Villingen, Germany
- Shatin, Hong Kong
- India (5):
  - Haryāna
  - New Dehli
  - New Delhi
  - Rajasthan
  - Vizag
- Kuala Lumpur, Malaysia
- Tal-Qroqq, Malta
- Lahore, Pakistan
- Poland (3):
  - Bydgoszcz
  - Krakow
  - Zabreze
- San Juan, Puerto Rico
- Romania (2):
  - Brasov
  - Bucharest
- Novena, Singapore
- Taiwan (2):
  - Taichung
  - Taipei
- Bangkok, Thailand

RESULTS

PARTICIPANT FLOW:
Groups:
- Attain Family Left Heart Lead: Subjects who underwent an Attain Family lead implant after either an Attain Family catheter attempt or any catheter model attempt
Period: Overall Study
Arm/Group | Attain Family Left Heart Lead
Started | 2014 (Total number of subjects enrolled)
Attain Family Study System Attempt | 1917 (Total number of subjects with an Attain Family lead attempt after an Attain Family catheter attempt)
Completed | 1802 (Total number of subjects with successful Attain Family lead using Attain Family catheter)
Not Completed | 212

BASELINE CHARACTERISTICS:
Groups:
- Attain Family Lead: Subjects who underwent an Attain Family lead implant after either an Attain Family catheter attempt or any catheter model attempt
Arm/Group | Attain Family Lead
Number analyzed (Participants) | 2014
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 661
  >=65 years | 1353
Age Continuous [Mean (Standard Deviation); unit: years] | 69.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 576
  Male | 1438
Region of Enrollment [Number; unit: participants]
  United States | 1648
  Taiwan | 30
  Hong Kong | 7
  Pakistan | 11
  Thailand | 4
  Malta | 8
  India | 79
  France | 83
  Canada | 15
  Puerto Rico | 35
  Malaysia | 12
  Poland | 22
  Singapore | 3
  Romania | 5
  Germany | 6
  China | 46

OUTCOME MEASURES:

1. Primary Outcome: Subjects Successfully Implanted With an Attain Family Left-heart Lead Using an Attain Family Delivery Catheter
Description: Implant success was defined as final successful placement of the Attain Family left-heart lead in the coronary vein branches utilizing the Attain Family of delivery catheters.
Time Frame: Implant
Measure: Number; unit: participants
Groups:
- Attain Family Lead and Catheter Attempt: Subjects who were attempted with an Attain Family left-heart lead after successful coronary sinus (CS) cannulation with an Attain Family catheter were included in this analysis as well as subjects who had unsuccessful CS cannulation with an Attain Family delivery catheter.
Arm/Group | Attain Family Lead and Catheter Attempt
Number analyzed (Participants) | 1917
participants | 1802 [.929 to .950]
Statistical Analysis 1: Comparison: Attain Family Lead and Catheter Attempt; Test type: Superiority or Other; One sample proportion = .940, 95% CI 2-sided [.929 to .951]

2. Primary Outcome: Subjects Without a Left-heart Lead and Delivery Catheter Related Complication
Description: A left-heart lead and delivery related complication was defined as a complication, an adverse event that resulted in death, any termination of significant device function or invasive intervention, that resulted from the presence of or performance (intended or otherwise) of the Medtronic left-heart lead or Attain Family of delivery catheters. All adverse events were adjudicated by an Adverse Event Advisory Committee (AEAC).
Time Frame: Implant to 3 months
Measure: Number; unit: participants
Groups:
- Attain Family Lead Attempt, Any Catheter: Subjects who were attempted with Attain Family delivery catheters or Attain Family left-heart leads were included in this analysis.
Arm/Group | Attain Family Lead Attempt, Any Catheter
Number analyzed (Participants) | 1944
participants | 1895
Statistical Analysis 1: Comparison: Attain Family Lead Attempt, Any Catheter; Test type: Superiority or Other; One sample proportion = .974, 95% CI 2-sided [.965 to .980]

ADVERSE EVENTS:
Time Frame: Implant to 3 month visit.
Description: All new and/or worsening adverse events related to the left heart leads and left heart delivery catheters were collected through the 3 month visit. Event collection began when the subject was enrolled in the study and underwent a left-heart lead implant attempt.
Groups:
- Attain Family Lead: All new and/or worsening adverse events related to the left-heart leads and left-heart lead delivery catheters were collected through the 3 month visit. Event collection started once the subject enrolled in the study and underwent a left-heart lead implant attempt.
Arm/Group | Attain Family Lead
Serious Adverse Events (participants affected / at risk) | 55/2014
Other Adverse Events (participants affected / at risk) | 0/2014
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Attain Family Lead (N=2014)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Device capturing issue (Injury, poisoning and procedural complications) | 2 (2)
Device connection issue (Injury, poisoning and procedural complications) | 1 (1)
Device dislocation (Injury, poisoning and procedural complications) | 29 (29)
Device pacing issue (Injury, poisoning and procedural complications) | 2 (2)
Device stimulation issue (Injury, poisoning and procedural complications) | 8 (8)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Implant site infection (Infections and infestations) | 4 (4)
Implant site irritation (Injury, poisoning and procedural complications) | 1 (1)
Pericardial haemorrhage (Cardiac disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sudden cardiac death (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No